CLINICAL TRIAL: NCT02633787
Title: Persistence of Bactericidal Antibodies in Adults Who Received a Booster Dose of Menactra® Approximately Four Years Earlier
Brief Title: Persistence of Bactericidal Antibodies in Adults Who Received a Booster Dose of Menactra® Approximately 4 Years Earlier
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTA00093; U1111-1161-3151 (Other: WHO)
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; Menactra®
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants received a booster dose of Menactra vaccine approximately four years earlier
  Interventions: Biological: Meningococcal (Groups A, C, Y, and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal (Groups A, C, Y, and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — No vaccine will be administered in this trial
  Other Names: Menactra®

SUMMARY:
The aim of this study is to provide information on the persistence of bactericidal antibodies following Menactra booster vaccination in study MTA77 ( NCT01442675).

Objective:

* To evaluate the persistence of antibody responses (determined by a serum bactericidal assay using human complement (SBA-HC)) approximately 4 years after the administration of a booster dose of Menactra vaccine in trial MTA77

DETAILED DESCRIPTION:
All eligible subjects will provide 1 blood sample at Visit 1. The duration of each subject's participation in the trial will be the duration of 1 visit (for enrollment and blood draw)

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years on the day of inclusion
* Received booster dose of Menactra vaccine in trial MTA77
* Informed consent form has been signed and dated
* Able to attend the scheduled visit and to comply with all trial procedures.

Exclusion Criteria:

* Participation at the time of trial enrollment (or in the 4 weeks preceding trial enrollment) in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any meningococcal vaccine, including serogroup B meningococcal vaccine, after receipt of the booster dose of Menactra vaccine administered in trial MTA77
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically
* Bleeding disorder, thrombocytopenia, or receipt of anticoagulants contraindicating venipuncture at the discretion of the Investigator
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Any illness that, in the opinion of the Investigator, might interfere with trial conduct or trial results
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the blood draw. (A prospective subject should not be included in the trial until 72 hours has passed.)
* Identified as an Investigator or employee of the Investigator or trial center with direct involvement in the proposed trial, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (4):
- United States (4):
  - Bardstown, Kentucky
  - Woburn, Massachusetts
  - Niles, Michigan
  - Layton, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 15 December 2015 to 28 December 2015 at 4 clinic sites in the United States.
Pre-assignment Details: A total of 110 participants who met all inclusion and none of the exclusion criteria were enrolled; 109 participants completed the trial.
Groups:
- All Subjects; Menactra Vaccine: Participants who received a booster dose of Menactra vaccine in trial MTA77 and were enrolled in MTA00093.
Period: Overall Study
Arm/Group | All Subjects; Menactra Vaccine
Started | 110
Completed | 109
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects; Menactra Vaccine: Participants who received a booster dose of Menactra vaccine in trial MTA77 (NCT01442675) and were enrolled in MTA00093.
Arm/Group | All Subjects; Menactra Vaccine
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 110
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.2 (3.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 49
Region of Enrollment [Number; unit: Participants]
  United States | 110

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Meningococcal Antibody Titers ≥ 1:4 Before, 28 Days After, and Approximately Four Years Following Menactra Vaccine Booster Vaccination.
Description: Anti-meningococcal antibody titers for serogroups A, C, Y, and W-135 were measured using a serum bactericidal assay with human complement.
Time Frame: Pre-booster vaccination, 28 days, and 4 years post-booster vaccination
Population: Anti-meningococcal antibody titers were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | All Subjects; Menactra Vaccine
Number analyzed (Participants) | 109
Percentage of participants
  Serogroup A; Pre-booster (N=108) | 88.0
  Serogroup A; 28 days post-booster (N=109) | 100.0
  Serogroup A; 4 years post-booster (N=109) | 98.2
  Serogroup C; Pre-booster (N=108) | 67.6
  Serogroup C; 28 days post-booster (N=109) | 100.0
  Serogroup C; 4 years post-booster (N=109) | 89.9
  Serogroup Y; Pre-booster (N=108) | 57.4
  Serogroup Y; 28 days post-booster (N=109) | 100.0
  Serogroup Y; 4 years post-booster (N=109) | 98.2
  Serogroup W-135; Pre-booster (N=108) | 83.3
  Serogroup W-135; 28 days post-booster (N=109) | 100.0
  Serogroup W-135; 4 years post-booster (N=109) | 97.2

2. Primary Outcome: Percentage of Participants With Meningococcal Antibody Titers ≥ 1:8 Before, 28 Days After, and Approximately Four Years Following Menactra Vaccine Booster Vaccination
Description: as for outcome 1
Time Frame: Pre-booster vaccination, 28 days and 4 years post-booster vaccination
Population: Anti-meningococcal antibody titers were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | All Subjects; Menactra Vaccine
Number analyzed (Participants) | 109
Percentage of participants
  Serogroup A; Pre-booster (N=108) | 67.6
  Serogroup A; 28 days post-booster (N=109) | 100.0
  Serogroup A; 4 years post-booster (N=109) | 94.5
  Serogroup C; Pre-booster (N=108) | 53.7
  Serogroup C; 28 days post-booster (N=109) | 100.0
  Serogroup C; 4 years post-booster (N=109) | 81.7
  Serogroup Y; Pre-booster (N=108) | 46.3
  Serogroup Y; 28 days post-booster (N=109) | 100.0
  Serogroup Y; 4 years post-booster (N=109) | 97.2
  Serogroup W-135; Pre-booster (N=108) | 72.2
  Serogroup W-135; 28 days post-booster (N=109) | 100.0
  Serogroup W-135; 4 years post-booster (N=109) | 95.4

3. Primary Outcome: Geometric Mean Titers of Meningococcal Antibodies Before, 28 Days After, and Approximately Four Years Following Menactra Vaccine Booster Vaccination
Description: as for outcome 1
Time Frame: Pre-booster, 28 Days and 4 years post-booster vaccination
Population: Anti-meningococcal antibody titers were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | All Subjects; Menactra Vaccine
Number analyzed (Participants) | 109
Titers (1/dilution)
  Serogroup A; Pre-booster (N=108) | 9.33 [7.7 to 11.3]
  Serogroup A; 28 days post-booster (N=109) | 460 [348.4 to 606.2]
  Serogroup A; 4 years post-booster (N=109) | 57.8 [44.2 to 75.6]
  Serogroup C; Pre-booster (N=108) | 11.2 [8.0 to 15.8]
  Serogroup C; 28 days post-booster (N=109) | 1224 [930.1 to 1609.6]
  Serogroup C; 4 years post-booster (N=109) | 54.6 [36.8 to 81.0]
  Serogroup Y; Pre-booster (N=108) | 7.50 [5.6 to 10.0]
  Serogroup Y; 28 days post-booster (N=109) | 1650 [1301.2 to 2091.8]
  Serogroup Y; 4 years post-booster (N=109) | 120 [88.9 to 162.3]
  Serogroup W-135; Pre-booster (N=108) | 13.4 [10.4 to 17.3]
  Serogroup W-135; 28 days post-booster (N=109) | 1170 [881.5 to 1553.8]
  Serogroup W-135; 4 years post-booster (N=109) | 93.1 [69.4 to 125.0]

ADVERSE EVENTS:
Time Frame: Monitoring of safety events was limited to serious adverse events considered related to study procedures (i.e., collection of the blood sample).
Description: As no vaccine was administered in this trial, monitoring of safety events was limited to serious adverse events considered related to study procedures (i.e., collection of the blood sample). No safety events were reported. This was an immunogenicity assessment involving participants of an earlier study MTA77 (NCT01442675).
Arm/Group | All Subjects; Menactra Vaccine
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.